CLINICAL TRIAL: NCT06006637
Title: Integrated Platform for Measuring and Reducing Symptoms of Autism Spectrum Disorder
Acronym: IPMR ASD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: JelikaLite LLC (Industry); Mt. Sinai School of Medicine, New York, New York (Unknown); MetroEHS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2041726; 111111 (Other Grant/Funding Number: FUZEhub)
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2024-12

CONDITIONS: Autism Spectrum Disorder
Keywords: Transcranial photobiomodulation; Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: This is a Randomized, Sham-controlled, Double Blind, Mixed-Design study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants and their caregivers will be held blind to group assignment. The PI will also remain blind to participant group assignment and conduct the pre- and post-assessment batteries (i.e., CARS-2, SRS, and CGI-I). Two clinical research assistants and co-investigator, will randomly assign participants to groups and have knowledge of their assignment. A third research assistant will also be held blind to group assignment and complete weekly interviews with caregivers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- CognilumTM (Experimental): During the study participants will be wear the transcranial photobiomodulation device Cognilum. The device will administer the stimulation of near infrared light (830nm) to specific areas of the child's brain.
  Interventions: Device: Cognilum TM: Light Treatment Condition
- Sham control (Sham Comparator): During the study participants will wear the transcranial photobiomodulation device. The device will not be turned on and therefore no brain stimulation with near infrared light (830nm) will be provided.
  Interventions: Device: Cognilum TM: Light Treatment Condition

INTERVENTIONS:
Device: Cognilum TM: Light Treatment Condition — The children will wear the CognilumTM device for approximately 10 minutes at a time, twice a week, for a period of 10 weeks.

SUMMARY:
This study will consist of a randomized, double-blind, sham-controlled clinical trial at SUNY Upstate Medical University and Mt. Sinai Medical Center with 80 autistic children evaluating the effects of transcranial photobiomodulation (tPBM) on multiple clinically validated scales.

DETAILED DESCRIPTION:
The proposed intervention will noninvasively deliver near infra-red (NIR) light - transcranial Photobiomodulation (tPBM) - to the brains of autistic children. The NIR light is delivered to specific brain areas by Cognilum, a wearable device developed by Jelikalite. The Cognilum system is a non-invasive headband medical device specifically designed to safely and comfortably deliver tPBM to autistic children. Cognilum has been designated as a non-significant risk breakthrough device by the Food and Drug Administration. This study will consist of a randomized, double-blind, sham-controlled clinical trial at SUNY Upstate Medical University and Mt. Sinai with 80 autistic children using Cognilium device and measuring the impact using multiple clinically validated scales.

Hypothesis 1: Significant reduction of average Childhood Autism Rating Scores (CARS; before and after treatment comparison) in the active group compared to sham-control group.

Hypothesis 2: Significant change in average scores (before and after treatment comparison) on the Social Responsiveness Scale (SRS), and Clinical Global Impression - Improvement (CGI-I) scale in the active group compared to sham control group.

ELIGIBILITY:
Inclusion Criteria:

* Ages 2 - 8
* Autism spectrum disorder diagnosis
* CARS-2 score of 30 - 45

Exclusion Criteria:

* CARS scores less than 30 or over 45.
* Taking psychotropic medications.
* Having skin lesions on scalp
* Having history of seizures
* Having history of abnormal EEG
* Being a relative of the PI or a researcher
* Having implanted devices (including cochlear implants).

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Childhood Autism Rating Scale, Second edition | 10 weeks
  Psychometrically sound measure for identifying children with autism and their symptom severity through quantifiable ratings based on direct observation. Raw scores may range from 15 to 60, which are then converted to T-scores. Higher scores indicate greater severity.

SECONDARY OUTCOMES:
Social Responsiveness Scale, Second Edition | 10 weeks
  Psychometrically sound measure for identifying the presence and severity of social impairment within the autism spectrum and differentiates it from that which occurs in other disorders. Raw scores may range from 65 to 260, which are then converted to T-scores. Higher scores indicate greater severity.
Clinical Global Impressions Scale | 10 weeks
  A well-established, brief assessment of the clinician's view of the patient's global functioning prior to and after initiating intervention. Ratings range from 1 (Normal) to 7 (Among the most severe).

OTHER OUTCOMES:
Clinical Interviews | 10 weeks
  Caregiver interviews obtaining information on the participant's functioning.
Aberrant Behavior Checklist | 10 weeks
  Behavior assessment
Repetitive Behavior Scale | 10 weeks
  Assessment of restricted and repetetive behaviors
Sensory Profile Caregiver Questionnaire -- Second Edition | 10 weeks
  Assessment of sensory needs

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Mt. Sinai Medical Center, New York, New York
  - Golisano Center for Special Needs, Syracuse, New York

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be available to other researchers